CLINICAL TRIAL: NCT01858480
Title: Randomized, Double-Blind, Placebo-Controlled Study To Evaluate D-Ribose For The Treatment Of Congestive Heart Failure
Brief Title: Study To Evaluate D-Ribose For The Treatment of Congestive Heart Failure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow enrollment
Sponsor: RiboCor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC 04C 010
Record Dates: First submitted 2013-05-09; First posted 2013-05-21 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Congestive Heart Failure
Keywords: CHF
MeSH Terms: conditions — Heart Failure | interventions — Ribose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-ribose (Active Comparator): D-ribose administered via peripheral intravenous for 24 hours followed by oral D ribose dosing for 3 months versus placebo in subjects with CHF who have been stabilized following hospitalization for acute decompensation.
  Interventions: Drug: D-ribose
- Placebo (Placebo Comparator): Placebo dosage form designed to mock active.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: D-ribose — D-ribose powder for oral solution and D-ribose for injection.
  Other Names: ribose
  Arms: D-ribose
Other: Placebo — Placebo dosage form designed to mock active.
  Arms: Placebo

SUMMARY:
To evaluate the safety and to determine the efficacy of D-ribose for the treatment of congestive heart failure (CHF) in subjects who have been stabilized following hospitalization with acute decompensation.

DETAILED DESCRIPTION:
This is a phase IIa, randomized, double-blind, placebo-controlled, multi-center study of D-ribose administered via peripheral intravenous line for 24 hours to stabilized hospitalized patients following standard of care treatment for acute decompensation of CHF, followed by oral dosing of D-ribose three times a daily through the remainder of the inpatient hospital stay and outpatient period of 3 months. Subjects will complete Pretreatment Screening procedures only after the Investigator has established that they have met the pre-specified criteria for stabilization of heart failure, and be randomized to treatment no more than 7 days after admission to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent and Health Insurance Portability and Accountability Act authorization, as applicable;
* symptomatic heart failure (NYHA Class II, III or IV) ≥ 30 days prior to current acute decompensation episode;
* ≥2 of the following signs of acute decompensation: jugular venous distension, rales, dyspnea, and ≥ 1+ pedal edema;
* admitted to the hospital ≤ 36 hours after initial evaluation;
* discontinued from IV inotropic support ≥ 48 hours prior to Screening;
* initiated Screening when subject has met the following criteria for stabilization:
* exacerbating factors addressed;
* near optimal volume status;
* transition from IV to oral diuretic completed;
* near optimal pharmacologic therapy achieved or intolerance documented;
* completed Screening procedures and been randomized to treatment ≤ 7 days after hospital admission;
* LVEF ≤ 35% ≤ 12 months prior to Screening.
* if female, ≥ 2 years post-menopausal, surgically sterile, or practicing effective contraception;
* if female, non-lactating, and if of child-bearing potential, has negative pregnancy test result at Screening;
* willing to abstain from ribose-containing products during study.

Exclusion Criteria:

* significant medical condition(s) which, in Investigator's judgment, could compromise subject's welfare or confound study results;
* significant hepatic, renal, or hematologic disorder/dysfunction beyond that expected from CHF alone;
* Creatinine Clearance <30.0 mL/min at Screening;
* serum potassium level <3.5 milliequivalent per liter or >5.7 milliequivalent per liter, or a serum sodium level <130 milliequivalent per liter at Screening;
* systolic arterial blood pressure <90 mm Hg at Screening;
* received ultrafiltration during current admission;
* cardiac surgery ≤ 60 days prior to Screening, except for percutaneous intervention;
* planned revascularization procedures, electrophysiologic device or cardiac mechanical support implantation, cardiac transplantation, or other cardiac surgery ≤ 90 days after study enrollment;
* functional mitral valve regurgitation > moderate severity;
* aortic regurgitation of at least moderate severity;
* hemodynamically significant primary cardiac valvular disease;
* myocardial infarction ≤ 30 days prior to Screening;
* Acute Coronary Syndrome ≤ 30 days prior to Screening;
* known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunt;
* sustained ventricular tachycardia or ventricular fibrillation ≤ 30 days prior to Screening, unless automatic implantable cardioverter defibrillator is present;
* atrial fibrillation within the past year;
* CHF related to tachyarrhythmias or bradyarrhythmias;
* CHF due to uncorrected thyroid disease, active myocarditis, or known amyloid cardiomyopathy;
* angina at rest or with slight exertion and/or unstable angina;
* diagnosed with hypertrophic cardiomyopathy;
* cerebrovascular accident ≤ 6 months prior to Screening;
* cardiogenic shock at any time from initial evaluation to randomization;
* on cardiac mechanical support;
* biventricular pacer placement ≤ 60 days prior to Screening or needed pacemaker placement during the current admission;
* refractory, end-stage heart failure;
* type I or type II diabetes;
* history of pancreatitis;
* current systemic infection;
* urinary tract obstruction;
* morbidly obese (weight > 159 kg [350 lbs] or BMI >42 kg/m2);
* active malignancy at Screening. [Treatment for basal cell or stage 1 squamous cell carcinoma, or cervical carcinoma in situ allowed];
* terminally ill or has moribund condition;
* history of irritable bowel syndrome, inflammatory bowel disease, ischemic colitis, vascular intestinal atherosclerosis, previous bowel resection, impaction, or similar gastrointestinal conditions;
* currently taking Kayexalate® (sodium polystyrene sulfonate);
* allergic reaction to Optison™ or Definity® or any of their components.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF), measured by transthoracic 2-D echocardiography with contrast | LVEF (by 2-D echocardiography): Change from Baseline to Month 3
  Efficacy Analyses: The primary efficacy analysis will be performed by comparison of active versus placebo treatment groups. Summary statistics, including means and standard deviations, will be provided. Analysis of covariance will be used to analyze the on-treatment LVEF scores with the pre-treatment LVEF score serving as the covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson S Colucci, MD, Study Chair — Boston University
Locations (24):
- United States (20):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Novo Research, Inc., Modesto, California
  - Olive View-UCLA- Medical Center, Sylmar, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Southeast Regional Research Group, Columbus, Georgia
  - Mercer University - Mercer Medicine, Macon, Georgia
  - Medical Consultants PC, Muncie, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - MedPharmics, Kenner, Louisiana
  - Androscoggin Cardiology Associates / dba Maine Research Associates, Auburn, Maine
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Genesys Regional Medical Ctr, Grand Blanc, Michigan
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Michael DeBakey VAMC, Houston, Texas
- Canada (4):
  - St. Michael's Hospital, Toronto, Ontario
  - Chum Hotel Dieu, Montreal, Quebec
  - Montreal General Hospital / MUHC, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
Study terminated due to slow enrollment